CLINICAL TRIAL: NCT03947905
Title: Comparison of Virtual to Physical Health Assessments and Treatment Plans for Patients Presenting for Initial Vascular Clinic Visits
Brief Title: Virtual and Physical Health Assessments and Treatment Plans
Acronym: VHAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CAMC Health System (Other)
Collaborators: Sarah & Pauline Maier Foundation, Inc. (Other); WVCTSI (Unknown)
Responsible Party: Principal Investigator, Albeir Mousa, Principal Investigator, CAMC Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-558
Record Dates: First submitted 2019-04-12; First posted 2019-05-13 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Vascular Diseases
Keywords: Vascular; Clinic visit; Tele-health
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Single arm crossover design where all participants receive both types of visits (Virtual and Physical visits).
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type of visit (Experimental): Single arm, non-randomized crossover design. All patients will receive both types of visits virtual and physical, and after assessments are made, participants will be classified by physicians into low, moderate or high risk for intervention.
  Interventions: Procedure: Virtual visit

INTERVENTIONS:
Procedure: Virtual visit — Type of visit
  Other Names: Physical visit

SUMMARY:
The aim of the current study is to compare virtual clinic visits (i.e., real-time, face-to-face visits conducted over the internet with tablet devices) to actual physical clinic visits. After both types of visits (virtual versus physical) physicians will be asked to classify patients into low, moderate or high risk for a vascular intervention. It is hypothesized that there will be good agreement between classifications made after the virtual visits as compared to those made after physical visits. That is, virtual visit classifications will be as good as those made after physical visits.

DETAILED DESCRIPTION:
Patient dissatisfaction can increase because of the complexities associated with navigating modern health care systems. It is easy to speculate that some of this dissatisfaction is associated with travel, wait times and other issues that arise during routine clinic visits. The authors of recent studies have demonstrated that it is possible and feasible to conduct many routine visits remotely. It is our belief that virtual health assessments and treatment plans (VHAT) conducted remotely can be as effective, perhaps be more efficient and increase patient satisfaction when compared to regular physical health assessments and treatment plans (PHAT). Physicians want to provide optimal health care; however, in geographically isolated areas such as some locations in West Virginia that can be a challenge. It seems reasonable to believe that monitoring patients with telehealth technology, collecting on-going real time data and conducting VHAT can provide high quality health care for patients. It can also help to classify health risk, increase patient and medical staff satisfaction, decrease staff time for visits, while at the same time increase the efficiency of the follow-up process. The investigators plan to compare the physician assessments and future treatment plans made using VHAT to those made after PHAT. It is believed that VHAT assessments will be in agreement with those made with PHAT.

ELIGIBILITY:
Inclusion Criteria:

-Patients referred to and scheduled for an initial visit at our Vascular Center of Excellence (VCOE).

Exclusion Criteria:

* Patients that are deemed urgent cases by the VCOE, and scheduled within two weeks for the initial clinic visit.
* Patients who are scheduled to have the placement of an arteriovenous (AV) fistula at the time of the initial clinic visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Categorization of physician treatment plans. (Physicians will classify treatment plans as low, moderate or high need for vascular intervention) | 1 week
  Comparison of virtual visit treatment plans to physical treatment plans. After assessments, physicians will classify patients' treatment plans into low (treat medically), moderate (vascular intervention in the future, but not immediately) or high (needs immediately, within 2 weeks). The distribution of low, moderate and high among the two types of visits (Virtual and Physical) will be compared.

SECONDARY OUTCOMES:
Patient satisfaction | 1 week
  Comparison of patient satisfaction after virtual and physical visits. Satisfaction will be measured by two survey questions based on a 1 to 5 Likert scale.

IPD SHARING:
Plan to Share IPD: No